CLINICAL TRIAL: NCT06663228
Title: Rapid Histologic Assessment for Stereotactic Breast Biopsy: Enhancing Early Detection With Miniature Mass Spectrometry and AI
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202405152RINB
Record Dates: First submitted 2024-07-15; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast biopsy; miniature mass spectrometry; artificial intelligence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- breast MMS
  Interventions: Diagnostic Test: MMS

INTERVENTIONS:
Diagnostic Test: MMS — miniature mass spectrometry with AI assistance

SUMMARY:
Breast cancer is the leading cancer among Taiwanese women, and it is the second leading cause of cancer-related deaths in women. The five-year survival rate for early-stage breast cancer (Stage 0 to II) is over 90%, significantly better than the survival rates for Stage III and Stage IV breast cancer, which are approximately 70% and 25%, respectively. As a result, breast cancer screening and early diagnosis have always been of great importance. Breast cancer screening relies on imaging examinations, and the diagnosis depends on imaging-guided tissue confirmation.

However, when a patient undergoes stereotactic breast biopsy due to suspicious lesions found in mammography, they typically have to wait about a week to receive the pathology results to determine whether the lesion is benign or malignant. For the patient, this waiting period can be agonizing, and for clinicians, earlier knowledge of pathology results would facilitate prompt staging evaluation and treatment planning for cancer.

The investigators use a special technique-paper spray ionization miniature mass spectrometry (PSI-MMS). According to preliminary research, with the assistance of AI, the miniature mass spectrometer can detect the benign or malignant nature of breast tissue within minutes and with decent accuracy. The investigators hope to continue research to further improve accuracy to meet clinical needs and aspire to have the opportunity to apply the miniature mass spectrometer to rapidly differentiate the molecular subtypes of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Those who come for receiving vacuum-assisted stereotactic breast biopsy

Exclusion Criteria:

* Those who cannot or are unwilling to sign the informed consent.

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females with abnormal mammography findings, that were categoried as ACR BI-RADS 4 or 5, come for vacuum-assisted stereotactic breast biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-07-04 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
breast cancer | July 2024 to July 2025
  PATHOLOGICAL DIAGNOSIS To prove the biopsy specimen to be malignant or benign.

CONTACTS AND LOCATIONS:
Locations (1):
- Jo-Yu Chen, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No